CLINICAL TRIAL: NCT06170398
Title: Interest of Electro-physiological Findings in the Assessment of Symptoms Severity in Superior Semi-circular Canal Dehiscence Syndrome
Brief Title: Electro-physiological Findings and Symptoms Severity in Superior Canal Dehiscence
Acronym: INTEX-DEHI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC31/22/0322; 2023-A01856-39 (Other: ID-RCB)
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Superior Semicircular Canal Dehiscence
Keywords: Superior semi-circular canal dehiscence; Minor syndrome; Pulsatile tinnitus; Autophony Tullio phenomenon
MeSH Terms: conditions — Semicircular Canal Dehiscence; Tinnitus | interventions — Audiometry, Evoked Response; Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Other): Electrophysiological tests
  Interventions: Diagnostic Test: Wideband tympanometry; Diagnostic Test: Electrocochleography; Diagnostic Test: Vestibular Evoked Myogenic potentials

INTERVENTIONS:
Diagnostic Test: Wideband tympanometry — Wideband tympanometry
Diagnostic Test: Electrocochleography — Electrocochleography
Diagnostic Test: Vestibular Evoked Myogenic potentials — Vestibular Evoked Myogenic potentials

SUMMARY:
This research aims at assessing the validity of three different electro-physiological tests (Vestibular Evoked Myogenic Potentials, WideBand Tympanometry, Electrocochleography) used in the investigation of the symptoms severity in the case of superior semi-circular canal dehiscence syndrome.

DETAILED DESCRIPTION:
Superior semi-circular canal dehiscence (SCD) syndrome can associate several cochlear and vestibular symptoms. Recent systematic reviews identified pulsatile tinnitus, autophony, sound-induced and pressure-induced vertigo as most specific signs of SCD. These signs are rarely all present and the symptomatology remains highly variable from a patient to another, with frequent though less evocative symptoms such as dizziness or ear pressure. A surgical treatment may be proposed when the symptoms become significantly incapacitating. Unfortunately to date, there is no objective marker of this severity and all surgical decisions rely on the importance of patients' complaints. High Resolution Computed Tomography (HRCT) of the temporal bone can confirm the diagnosis. Electro-physiological investigations such as Vestibular Evoked Myogenic potentials (VEMPs) have also been extensively described in the diagnosis of SCD but they have been reported as independent from the symptoms severity. Wideband tympanometry (WBT) and Electrocochleography (EcoG) have only been studied in few reports but the latter appears as a promising tool in the assessment of the symptoms because it explores inner ear biomechanics, directly involved in the pathophysiology of this condition.

ELIGIBILITY:
Inclusion Criteria:

* confirmed unilateral SCD (using specific HRCT settings and reconstructions) with or without SCD symptoms
* if present, SCD symptoms should be stable
* patients understanding and reading french
* affiliated to social security.

Exclusion Criteria:

* bilateral confirmed SCD
* doubtful SCD
* other otologic or neurotologic condition that might mimick SCD symptomatology : middle ear conditions, Meniere disease, vestibular migraine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
EcoG validity - pulsatile tinnitus | 30 day
  the validity of EcoG will be assessed by the correlation between the alteration of the summating potential/action potential ratio and symptom severity (pulsatile tinnitus) assessed by a visual analogue scale (0 to 10)
EcoG validity - autophony | 30 day
  the validity of EcoG will be assessed by the correlation between the alteration of the summating potential/action potential ratio and symptom severity (autophony) assessed by a visual analogue scale (0 to 10)
EcoG validity - dizziness induced by loud sounds | 30 day
  the validity of EcoG will be assessed by the correlation between the alteration of the summating potential/action potential ratio and symptom severity (dizziness induced by loud sounds) assessed by a visual analogue scale (0 to 10)
EcoG validity - dizziness induced by pressure changes | 30 day
  the validity of EcoG will be assessed by the correlation between the alteration of the summating potential/action potential ratio and symptom severity (dizziness induced by pressure changes) assessed by a visual analogue scale (0 to 10)

CONTACTS AND LOCATIONS:
Overall Officials: Yohan GALLOIS, Dr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Legois Q, Giraudet F, Gallois Y, Lepage B, Ionescu E, Vellin JF, Franco-Vidal V, Kaderbay A, Vellin MJ; French Association of Superior Semicircular Canal Dehiscence syndrome; Marx M. INTerest of electrophysiological and functional EXploration in the evaluation of symptomatic impact of superior semicircular canal DEHIscence syndrome (INTEX-DEHI study): Study protocol for a reliability and validity study. PLoS One. 2025 Sep 18;20(9):e0331763. doi: 10.1371/journal.pone.0331763. eCollection 2025. PMID 40966240